CLINICAL TRIAL: NCT05090800
Title: Contrast Enhanced Ultrasound for Renal Obstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sapan Ambani, Associate Professor of Urology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00193843
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Kidney; Obstruction; Renal Obstruction
Keywords: ultrasound imaging; ultrasound contrast agents; kidney tissue; hydronephrosis
MeSH Terms: conditions — Bites and Stings; Hydronephrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Definity contrast agent (Experimental)
  Interventions: Drug: Definity contrast during ultrasound

INTERVENTIONS:
Drug: Definity contrast during ultrasound — Participants will undergo an ultrasound contrast evaluation of both kidneys. This will include placement of an intravenous (IV) catheter in a vein and the delivery of Definity ultrasound contrast agent through the IV. Imaging will be completed for each kidney. The proposed total dose for adult patients will not exceed 20 microliters/kilograms (kg). Each individual dose not to exceed 10 microliters/kg. At initiation of patient studies, the dose will start at 10 microliters/kg for the first injection and a second 10 microliters/kg dose to evaluate the contralateral kidney. However, if ultrasound findings in patient studies demonstrate a dose that is too high (unable to make accurate ultrasound assessment), the dose will be reduced.
  Other Names: Perflutren Lipid Microsphere

SUMMARY:
This research is studying Definity ultrasound contrast agent, which is already approved by the Food and Drug Administration (FDA) for the ultrasound evaluation of the liver and heart. This research will investigate the ability to use ultrasound imaging with ultrasound contrast agents to evaluate kidney obstruction.

Eligible participants that are enrolled will have two visits (one before and one after the planned surgery to relieve the kidney obstruction).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral renal obstruction confirmed by Nuclear Medicine MAG3 Dynamic Renal Scan (diuretic t (time) ½ >20 minutes)
* Obstructed kidney with differential function >15% confirmed by Nuclear Medicine Mercaptoacetyltriglycine (MAG3) Dynamic Renal Scan within less or equal (<=) 6 months from enrollment
* Patient has elected to move forward with pyeloplasty or proximal ureteroureterostomy to correct the obstruction

Exclusion Criteria:

* Solitary kidney
* Any abnormalities of contralateral collecting system (for example (e.g.) hydronephrosis, renal calculi, duplicated collecting system)
* Known vesicoureteral reflux
* Ureteral stent in place in the obstructive kidney
* Patients without a Nuclear Medicine MAG3 Dynamic Renal Scan
* Previous history of hypersensitivity to Ultrasound Contrast Agents or Definity (perflutren lipid microspheres))
* Previous sensitivity to polyethylene glycol
* Pregnant or breastfeeding females
* Body mass index (BMI) >=40 without prior ultrasound confirming ability to adequately visualize the kidneys (Elevated BMI is known to decrease ability to image the kidneys)
* Global renal function with a Glomerular Filtration Rate (GFR) <30 (chronic kidney disease Stage 4 & 5 excluded)
* Unstable cardiopulmonary conditions (acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, serious ventricular arrhythmias, presence of a cardiac shunt)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Time to peak (TTP) ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Peak intensity (PI) ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Mean transit time (MTT) ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Area under the curve (AUC) ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Ratio of plateau and peak intensity ultrasound Measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys

SECONDARY OUTCOMES:
Contrast arrival time (AT) ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Enhanced slope ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Fall time (FT) ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Time from peak to baseline (TPB) ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Final plateau intensity ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys
Initial intrarenal microcirculatory transmit time ultrasound measurements | Immediately after contrast injected (approximately 30 minutes)
  Differences in ultrasound contrast measurements between obstructed and normal kidneys

CONTACTS AND LOCATIONS:
Overall Officials: Sapan N Ambani, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No